CLINICAL TRIAL: NCT02489786
Title: A Prospective Randomized Study of Different Digoxin Treatment Regimens in Egyptian Hospital
Brief Title: A Prospective Study of Different Digoxin Treatment Regimens in Egyptian Hospital
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Atef ALShabasy, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (312)
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen 1 (Active Comparator): patient takes 0.25mg of digoxin daily except friday
  Interventions: Drug: patients take 0.25 mg of digoxin daily except friday
- Regimen 2 (Active Comparator): patient takes 0.25mg of digoxin daily except Thursday and Friday
  Interventions: Drug: patients take 0.25 mg of digoxin daily except thursday and friday
- Regimen 3 (Active Comparator): patient takes 0.125mg of digoxin daily
  Interventions: Drug: patients take 0.125 mg of digoxin daily
- Regimen 4 (Active Comparator): digoxin dose is calculated using Jusko-Koup method and given daily
  Interventions: Drug: digoxin dose is calculated using Jusko-Koup method and given daily

INTERVENTIONS:
Drug: patients take 0.25 mg of digoxin daily except friday
  Arms: Regimen 1
Drug: patients take 0.25 mg of digoxin daily except thursday and friday
  Arms: Regimen 2
Drug: patients take 0.125 mg of digoxin daily
  Arms: Regimen 3
Drug: digoxin dose is calculated using Jusko-Koup method and given daily
  Arms: Regimen 4

SUMMARY:
Digoxin is the primary cardiac glycoside in clinical use. Because of the narrow therapeutic index and risk of toxicity, therapeutic drug monitoring is highly recommended. In Egypt, most cardiologists give digoxin holiday for both atrial fibrillation and heart failure, it is not clear if the interrupted digoxin regimens are effective since serum digoxin concentrations might fall below the therapeutic range.

Objective: To evaluate and compare the digoxin serum concentration and patient's quality of life in the continuous versus interrupted digoxin dosing regimens.

DETAILED DESCRIPTION:
Digoxin is a cardiac glycoside prescribed in heart failure and certain supraventricular tachyarrhythmias. It exerts a positive inotropic, neurohormonal, and electro physiologic actions on the heart . For heart failure patients, the targeted steady state serum digoxin level is between 0.5 and 0.8 ng/ml . Ventricular rate control in atrial fibrillation patients will usually require higher digoxin steady state serum concentrations . However, serum digoxin level higher than 2 ng/ml is associated with increased incidence of adverse drug reactions and should be avoided . Because of inter and intra-patient variability, narrow therapeutic index, and risk of toxicity, digoxin doses are calculated based on the patient weight, renal status, indications and drug interactions. Due to substantial overlap between therapeutic and toxic levels of digoxin, therapeutic drug monitoring is a must especially in patients with deteriorating renal function and electrolyte disturbance. In Egypt, most cardiologists give a digoxin holiday for patients with atrial fibrillation and /or heart failure where patients skip the drug doses on Thursday and Friday or Friday only every week to avoid possible drug accumulation and toxicity. It is not clear if these interrupted digoxin regimens really offer safer alternative over the continuous dosing regimens without compromising the effectiveness. It is anticipated that plasma digoxin levels may fall below the therapeutic range during the holiday which may affect patient clinical status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation (AF)
* with or without congestive heart failure (CHF)
* taking digoxin tablets with or without holiday regimens

Exclusion Criteria:

* taking the following drugs concurrently: amiodarone, verapamil, quinidine and propafenone.
* diagnosed with thyroid disorders (hyperthyroidism & hypothyroidism).
* diagnosed with renal failure
* pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
measuring digoxin trough steady state plasma concentrations for the interrupted and continuous treatment regimens | 1 month

SECONDARY OUTCOMES:
evaluating patients quality of life using quality of life questionnaire for atrial fibrillation patients | 1 month
evaluating signs and symptoms of digoxin side effects and toxicity by using specific structured questions | 1 month